CLINICAL TRIAL: NCT05622513
Title: the Association Between Phthalate Esters and Childhood Obesity
Brief Title: Phthalate Esters and Childhood Obesity
Status: Completed | Type: Observational
Sponsor: Shenzhen Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Di Li, doctor, Shenzhen Center for Disease Control and Prevention
Other Study IDs: szCDC_3
Record Dates: First submitted 2022-11-13; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — urine sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: obesity / overweight children
- controls: normal weight children

SUMMARY:
Phthalate esters have been considered closely related with childhood obesity, but the existing studies revealed inconsistent results. This study was desigened to investigate the association between phthalate esters and childhood obesity in China.

DETAILED DESCRIPTION:
The physical activity, dietary intake and the levels of urine phthalate metabolites of children were detected, and the associations between these 3 factors and childhood obesity were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Children who were classified as normal, overweight and obesity based on age, gender and BMI.

Exclusion Criteria:

* The participants who were with endocrine disorders.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Students aged 6-8 years from monitoring schools in Shenzhen, China.
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
the levels of urine phthalate metabolites | 3 months
  9 phthalate metabolites (MMP, MEP, MnBP, MiBP, MEHP, MEOHP, MEHHP, MCEPP, MCMHP) in first morning urine sample of the participants were detected

REFERENCES:
- [Derived] Li D, Yao Y, Chen D, Wu Y, Liao Y, Zhou L. Phthalates, physical activity, and diet, which are the most strongly associated with obesity? A case-control study of Chinese children. Endocrine. 2023 Oct;82(1):69-77. doi: 10.1007/s12020-023-03465-w. Epub 2023 Aug 2. PMID 37532921